CLINICAL TRIAL: NCT03334721
Title: Gabapentin for Bipolar & Cannabis Use Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, James J. Prisciandaro, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 69905; R21DA04391701A1 (Other Grant/Funding Number: NIDA)
Record Dates: First submitted 2017-09-29; First posted 2017-11-07 (Actual); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Bipolar I Disorder; Bipolar II Disorder; Cannabis Use Disorder; Substance Use Disorders
MeSH Terms: conditions — Bipolar Disorder; Substance-Related Disorders | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin, Then Placebo Oral Capsule (Experimental): Week 1: 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Week 2: 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Interventions: Drug: Gabapentin; Drug: Placebo Oral Capsule
- Placebo Oral Capsule, Then Gabapentin (Experimental): Week 1: 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Week 2: 1-week condition will consist of an in-person study visit for assessment and dispensing of Gabapentin medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Interventions: Drug: Gabapentin; Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Gabapentin — 5 day trial of gabapentin with titration to 1,200mg
Drug: Placebo Oral Capsule — 5 day trial of matched placebo

SUMMARY:
The proposed 2-week, double-blind, crossover, proof of concept study aims to measure and manipulate core neurochemical (i.e., dysregulated brain GABA/glutamate homeostasis) and neurobehavioral (i.e., elevated impulsivity) dysfunctions characteristic of individuals with cannabis use disorder (CUD) and Bipolar Disorder (BD), using a medication that has been shown to increase cortical GABA (i.e., gabapentin) levels in past research, and to evaluate medication-related changes in response inhibition (go no-go) and cannabis cue reactivity functional Magnetic Resonance Imaging tasks, as well as cannabis use, mood symptoms (including anxiety and sleep), and impulsivity in individuals with CUD+BD.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is the Axis I condition most strongly associated with cannabis use disorder (CUD); there is a six-fold increase in the prevalence of CUD in individuals with BD relative to the general population. Individuals with co-occurring CUD and BD (CUD+BD) have substantially worse clinical outcomes than those with either BD or CUD alone. Response to mood stabilizing medications appears to be poor, yet little is known about optimal treatment for CUD+BD, as there have been no randomized medication trials for CUD+BD to date. Convergent evidence supports dysregulated brain γ-Aminobutyric acid (GABA)/glutamate homeostasis as a candidate target for pharmacological intervention in CUD+BD. Preclinical and clinical studies have demonstrated that CUD and BD are each associated with prefrontal GABA and glutamate disturbances and that impulsivity, a core neurobehavioral feature of both CUD and BD and a key Research Domain Criteria (RDoC) construct, is causally related to GABAergic/glutamatergic functioning. Gabapentin has been consistently shown in preclinical research to modulate GABA and glutamate transmission. In human Proton Magnetic Resonance Spectroscopy (1H-MRS) studies, both acute and chronic gabapentin dosing have been shown to increase brain GABA levels, however, few studies have investigated gabapentin effects on glutamate levels. Researchers propose that gabapentin may impact clinical outcomes in CUD+BD individuals both directly and indirectly through their impact on impulsivity.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-V criteria for Bipolar Disorder
* Meets DSM-V criteria for Cannabis Use Disorder
* Using at least one mood stabilizing medication

Exclusion Criteria:

* Serious medical or non-inclusionary psychiatric disease
* Concomitant use of benzodiazepine medications or any medications hazardous if taken with gabapentin
* History of clinically significant brain injury
* Presence of non-MRI safe material, or clinically significant claustrophobia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J Prisciandaro, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prisciandaro JJ, Mellick W, Squeglia LM, Hix S, Arnold L, Tolliver BK. Results from a randomized, double-blind, placebo-controlled, crossover, multimodal-MRI pilot study of gabapentin for co-occurring bipolar and cannabis use disorders. Addict Biol. 2022 Jan;27(1):e13085. doi: 10.1111/adb.13085. Epub 2021 Aug 14. PMID 34390300

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin, Then Placebo Oral Capsule: Week 1: 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Week 2: 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
  Placebo Oral Capsule: 5 day trial of matched placebo
- Placebo Oral Capsule, Then Gabapentin: Week 1: 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Week 2: 1-week condition will consist of an in-person study visit for assessment and dispensing of Gabapentin medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
  Placebo Oral Capsule: 5 day trial of matched placebo
Period: Overall Study
Arm/Group | Gabapentin, Then Placebo Oral Capsule | Placebo Oral Capsule, Then Gabapentin
Started | 12 | 11
Completed | 10 | 11
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — No longer met inclusion/exclusion criter | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gabapentin, Then Placebo Oral Capsule: Week 1: Gabapentin: 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Week 2: Placebo: 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
- Placebo Oral Capsule, Then Gabapentin: Week 1: Placebo: 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Week 2: Gabapentin: 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
- Total: Total of all reporting groups
Arm/Group | Gabapentin, Then Placebo Oral Capsule | Placebo Oral Capsule, Then Gabapentin | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 38.58 [25 to 63] | 35.45 [18 to 52] | 37.09 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Prefrontal GABA Concentrations Through Proton Magnetic Resonance Spectroscopy
Description: Concentrations of GABA, normalized to water and corrected for CSF%, in dorsal anterior cingulate measured via Proton Magnetic Resonance Spectroscopy.
Time Frame: Day 5 of each experimental condition
Population: Individuals with Bipolar Disorder and Cannabis Use Disorder
Measure: Mean (Standard Deviation); unit: Institutional Units
Groups:
- Gabapentin: Each 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (i.e., 1,200mg gabapentin) (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Gabapentin: 5 day trial of gabapentin with titration to 1,200mg
- Placebo Oral Capsule: Each 1-week condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), titration to maximum dose (Days 1-5), MRI (Day 5), and medication washout (Days 5-7).
  Placebo Oral Capsule: 5 day trial of matched placebo
Arm/Group | Gabapentin | Placebo Oral Capsule
Number analyzed (Participants) | 22 | 21
Institutional Units
  GABA (randomization order 1, gabapentin 1st): number analyzed (Participants) | 11 | 10
  GABA (randomization order 1, gabapentin 1st) | 2.625 (0.324) | 2.696 (0.313)
  GABA (randomization order 2, placebo 1st): number analyzed (Participants) | 11 | 11
  GABA (randomization order 2, placebo 1st) | 2.609 (0.290) | 2.720 (0.248)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo Oral Capsule; Test type: Superiority — Given the crossover design through which the data were collected, the statistical model also included a "Visit" (1 vs. 2) factor and a Visit by Treatment Condition interaction term. Analysis used Linear Mixed Modeling with Fixed Factors; p = 0.711, Mixed Models Analysis — Treatment Condition Factor (0 = Placebo, 1 = Gabapentin); df = 1, 20.183; Test III Tests of Fixed Effects (F) = 0.141; Given the crossover design through which the data were collected, the statistical model also included a "Visit" (1 vs. 2) factor and a Visit by Treatment Condition interaction term

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a total of 4 visits (Med 1, MRI 1, Med 2, MRI 2) for each participant; 2-weeks.
Description: Please note -23 participants took gabapentin but only 22 took placebo because one participant dropped out of the study prior to receiving the placebo oral capsule (this was a crossover study).
Arm/Group | Gabapentin | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 8/23 | 6/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=23) | Placebo Oral Capsule (N=22)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Increased Appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Memory Impairment (Nervous system disorders) | 1 (1) | 1 (1)
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT03334721/Prot_SAP_000.pdf